CLINICAL TRIAL: NCT05509569
Title: Specified Drug Use Surveillance of FIRAZYR Subcutaneous Injection 30mg Syringe for Pediatric Subjects With Hereditary Angioedema (All-Case Investigation)
Brief Title: A Survey of Icatibant in Pediatric Participants With Hereditary Angioedema
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-667-4003; jRCT2031220292 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant; Syringes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Icatibant: Participants will be recieved Icatibant 10 to 30 mg injection subcutaneously.
  Interventions: Drug: Icatibant

INTERVENTIONS:
Drug: Icatibant — Icatibant, 10 to 30 mg, Subcutaneous injection
  Other Names: FIRAZYR Subcutaneous Injection 30mg Syringe

SUMMARY:
This study is a survey in Japan of Icatibant subcutaneous injection 30 mg syringe used to treat children or teenagers with acute attacks of hereditary angioedema (HAE). The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects related from Icatibant subcutaneous injection 30 mg syringe and to check if Icatibant subcutaneous injection 30 mg syringe improves acute attacks of HAE.

During the study, pediatric participants with HAE will take Icatibant subcutaneous injection 30mg syringe according to their clinic's standard practice. The study doctors will check for side effects from Icatibant subcutaneous injection 30 mg syringe for 3 months.

ELIGIBILITY:
Inclusion Criteria:

- All participants with HAE who are 2 to <18 years of age, treated with Icatibant subcutaneous injection 30 mg syringe for the first time.

Exclusion Criteria:

- Participants who have been treated with Icatibant subcutaneous injection 30 mg syringe in clinical trials or transfer cases, and so on.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population of this survey are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least One Treatment-Emergent Adverse Events (TEAE) | Up to 3 Months

SECONDARY OUTCOMES:
Time from Onset of Seizure to Start of Treatment | Up to 3 Months
  Time from onset of seizure to the first drug administration will be assessed.
Time from First Drug Administration to Symptom Resolution | Up to 3 Months
  Time from the first drug administration to complete resolution of all symptoms of HAE will be assessed.
Duration of Seizure | Up to 3 Months
  The time from the start of the seizure to the disappearance of all symptoms will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/fcb2fbc9311e4e80